CLINICAL TRIAL: NCT02259335
Title: A Pilot Study on the Use of Extracorporeal CO2 Removal During the Weaning Process From Mechanical Ventilation
Brief Title: Weaning Form Mechanical Ventilation Using Extracorporeal CO2 Removal
Acronym: WeanPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Professor of Respiratory Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110/2014
Record Dates: First submitted 2014-10-04; First posted 2014-10-08 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Patients With Acute Hypercapnic Respiratory Failure
Keywords: weaning from mechanical ventilation; extracorporeal CO2 removal; post-extubation failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients under invasive ventilation (Experimental): those patients failing a T-piece trial beacuse of a PaCO2 rise>20% of baseline and/or a rapid shallow-breathing index >100 will be reconnected to the ventilator Two hours later they will repeat a T-piece trial after connection to the CO2 removal device
  Interventions: Device: Extracorporeal CO2 removal device

INTERVENTIONS:
Device: Extracorporeal CO2 removal device — A device able to remove CO2 using a dedicated device connected to the patient via a double lumen catheter inserted in the femoral vein
  Other Names: DeCap

SUMMARY:
Weaning from invasive mechanical ventilation is one of the major clinical problem especially ion those patients with a pre-existing chronic respiratory disease and chronic hypercpania.

The aim of this pilot feasibility and safety trial is to assess the possibility of shorten the duration of mechanical ventilation using a device able to remove CO2 and theoretically able to allow therefore the praecox extubation

DETAILED DESCRIPTION:
Weaning from invasive mechanical ventilation is one of the major clinical problem especially ion those patients with a pre-existing chronic respiratory disease and chronic hypercpania. Up to 60% of the ventilatory time is devoted in these patients to the process of weaning.

These patients very often fail several weaning attempt, when a T-piece trial method is used. In this case they are also very likely to require tracheotomy.

In this study we will enroll those still hypercapnic patients fitting the criteria of readiness to be wean (i.e. clinical stability, normal sensorium and good cough reflex) and failing a T-piece trail because of a rise in PaCO2 (>20% from baseline) and/or a rapid shallow breathing index (f/VT)> 100.

After the unsuccessful trial they will be reconnected to the ventilator and they will repeat hours later the same T-piece trial once the extracorporeal CO2 removal device (DeCap) will be connected via a double lumen catheter in the femoral vein.

The investigators aim to verify whether using the DeCap) the investigators will be able to avoid at the end of the T-piece trial the criteria of failure. If so, the patient will be extubated and DeCap will be continued when all of the following were achieved for at least 12 hours: respiratory rate less than 25 breaths/min; pH greater than 7.35; Paco2 less than 20% of the baseline value; and absence of use of the accessory muscles or paradoxical abdominal movements.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the criteria for readiness to be weaned (i.e. clinical stability, FiO2<50%, normal sensorium, body temperature < 38 and satisfactory cough reflex)
* Failing a T-piece trial after 1 hour or before for a rise in PaCO2>20% from baseline and with f/VT ratio >100

Exclusion Criteria:

* Patients NOT meeting the criteria for readiness to be weaned
* Patients succeeding a T-piece trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
passing a weaning trial using a T-piece method | 1 hour
  avoiding to reach the criteria of weaning failure
weaning success | 48 hours
  avoiding reintubation after removal of DeCap

SECONDARY OUTCOMES:
Physiological variables (i.e. Arterial Blood Gases, vitals and dyspnea) | 48 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - AOU Città della Salute e della Scienza di Torino, Molinette Hospital, Turin, Turin
  - San'Orsola Malpighi Hospital, Bologna ITALY, Bologna